CLINICAL TRIAL: NCT04831359
Title: Tissue Doppler Assessment of Right Ventricular Function in Newly Diagnosed Pediatric Cancer Patients Underwent Chemotherapy in South Egypt Cancer Institute
Brief Title: Tissue Doppler Assessment of Right Ventricle Function in Pediatrics Underwent Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham M Farghally, Resident, Assiut University
Other Study IDs: Tissue Doppler assesment
Record Dates: First submitted 2021-03-29; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Cancer Patients
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Doppler ultrasound — Tissue Doppler ultrasound on pediatric patients

SUMMARY:
Tissue Doppler assessment of right ventricular function in newly diagnosed pediatric cancer patients underwent chemotherapy in South Egypt Cancer Institute.

DETAILED DESCRIPTION:
The incidence of cancer is always increasing and it is predicted that the incidence will increase to 45% by 2030(1). The introduction of new chemotherapeutic agents significantly improved survival, but also revealed large spectrum of cardiotoxicity manifestations (2). There are many factors that increase the risk of cardiotoxicity caused by different chemotherapeutic agents, such as type of chemotherapy, cumulative dose, concomitant or previous radiotherapy, and comorbidities (3). Chemotherapeutic regimens which contain anthracyclines, cyclophosphamide, fluorouracil, cisplatin, taxanes and trastuzumab cause early and late cardiotoxicity (4).

The majority of published studies are focused on left ventricle dysfunction in patients receiving cardiotoxic chemotherapy. However, the right ventricle has been ignored for a long time and a little attention has been directed to show the effect of chemotherapy on right ventricle function. Right ventricle dysfunction is associated with increased morbidity and mortality in many cardiovascular diseases (5). The structure of cardiomyocytes and blood supply between the left and right ventricles are similar. Given the smaller mass and fewer myofibrils of right ventricle, chemotherapy may theoretically cause a more significant impact on it (6).

The right ventricle has a complex geometric shape which includes smooth muscular inflow, outflow and a trabecular apical region so echocardiographic assessment of right ventricle is difficult (7).

M-mode echocardiography, two-dimensional echocardiography, conventional Doppler echocardiography, and myocardial Doppler tissue imaging are all used to evaluate right ventricular function and provide accurate prognostic information especially when used in combination

ELIGIBILITY:
Inclusion Criteria:

* Patients of 1-18 years who are newly diagnosed to have cancer and will be referred to South Egypt cancer institute for receiving chemotherapy

Exclusion Criteria:

1. patients with left ventricular (EF) <50% before chemotherapy
2. Previous heart disease
3. Renal failure
4. significant valvular disease

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: - Patients of 1-18 years who are newly diagnosed to have cancer and will be referred to South Egypt cancer institute
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Effect of chemotherapy on right ventricular function | Baseline to 45 days
  The correlation between echocardiographic parameters of the RV, measured with transthoracic echocardiography before and after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith BD, Smith GL, Hurria A, Hortobagyi GN, Buchholz TA. Future of cancer incidence in the United States: burdens upon an aging, changing nation. J Clin Oncol. 2009 Jun 10;27(17):2758-65. doi: 10.1200/JCO.2008.20.8983. Epub 2009 Apr 29. PMID 19403886
- [Background] Dell'Italia LJ. The right ventricle: anatomy, physiology, and clinical importance. Curr Probl Cardiol. 1991 Oct;16(10):653-720. doi: 10.1016/0146-2806(91)90009-y. No abstract available. PMID 1748012
- [Background] Carver JR, Shapiro CL, Ng A, Jacobs L, Schwartz C, Virgo KS, Hagerty KL, Somerfield MR, Vaughn DJ; ASCO Cancer Survivorship Expert Panel. American Society of Clinical Oncology clinical evidence review on the ongoing care of adult cancer survivors: cardiac and pulmonary late effects. J Clin Oncol. 2007 Sep 1;25(25):3991-4008. doi: 10.1200/JCO.2007.10.9777. Epub 2007 Jun 18. PMID 17577017
- [Background] Surkova E, Muraru D, Iliceto S, Badano LP. The use of multimodality cardiovascular imaging to assess right ventricular size and function. Int J Cardiol. 2016 Jul 1;214:54-69. doi: 10.1016/j.ijcard.2016.03.074. Epub 2016 Mar 25. PMID 27057977
- [Background] Burgess MI, Bright-Thomas RJ, Ray SG. Echocardiographic evaluation of right ventricular function. Eur J Echocardiogr. 2002 Dec;3(4):252-62. No abstract available. PMID 12413440
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Koestenberger M, Ravekes W, Everett AD, Stueger HP, Heinzl B, Gamillscheg A, Cvirn G, Boysen A, Fandl A, Nagel B. Right ventricular function in infants, children and adolescents: reference values of the tricuspid annular plane systolic excursion (TAPSE) in 640 healthy patients and calculation of z score values. J Am Soc Echocardiogr. 2009 Jun;22(6):715-9. doi: 10.1016/j.echo.2009.03.026. Epub 2009 May 7. PMID 19423286